CLINICAL TRIAL: NCT07045090
Title: The Effect of Transcutaneous Electrical Acupoint Stimulation Combined With Transcutaneous Auricular Vagus Nerve Stimulation on Postoperative Delirium in Elderly Patients Undergoing Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Lulu Ji, Attending physician, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-K071-01
Record Dates: First submitted 2025-02-19; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Delirium
Keywords: Elderly patients; postoperative delirium; gastrointestinal surgery; Auricular vagus nerve stimulation; Transcutaneous electrical acupoint stimulation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Prior to induction of anaesthesia, patients in this group received transcutaneous electrical stimulation of acupuncture points for 30 min, followed by standardised anaesthesia.
  Interventions: Device: Transcutaneous electrical acupoint stimulation
- Group B (Experimental): Prior to induction of anaesthesia, patients in this group received transcutaneous electrical acupoint stimulation combined with auricular vagus nerve stimulation for a total of 30 min, followed by standardised anaesthesia.
  Interventions: Device: Transcutaneous electrical acupoint stimulation combined with auricular vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — Before induction of anaesthesia, electrodes were attached to selected acupoints and energised for 30 min, with the electrical stimulation parameter of dispersed dense wave (2/100 Hz), and the current intensity was based on the maximum current intensity that could be tolerated by the patient.
  Arms: Group A
Device: Transcutaneous electrical acupoint stimulation combined with auricular vagus nerve stimulation — Before anaesthesia induction, the electrodes were attached to the selected acupoints and energized for 30 min, with the electrical stimulation parameters of dispersed dense wave (2/100Hz), and the current intensity was based on the maximum current intensity that the patient could tolerate. At the same time, the left ear auricular region was stimulated with a fasciculus nerve stimulator, the electrical stimulation parameters were: pulse width of 250 μs, pulse frequency of 20Hz, every 30s on, 30s off, and then 30s on again, the current intensity was based on the maximum current intensity that the patient could tolerate, for 30min.
  Arms: Group B

SUMMARY:
The aim of this clinical trial is to study the effect of transcutaneous electrical acupoint stimulation combined with auricular vagus nerve stimulation on postoperative delirium in elderly patients undergoing gastrointestinal surgery. The study aims to answer the following main questions

1. whether it reduces the expression of inflammatory factors in the acute postoperative period
2. whether it can reduce the incidence of postoperative delirium

DETAILED DESCRIPTION:
Existing clinical studies have shown that TEAS has demonstrated value in preventing postoperative delirium (POD). Currently, taVNS is commonly used clinically to improve patients' cognitive dysfunction (POCD), and POD is often considered a precursor to the development of POCD. However, no one has yet used the two in combination, so this study aimed to combine the two to investigate their potential benefits in preventing POD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥65 years;
2. Body mass index (BMI) 18-30 kg/m²;
3. American Society of Anesthesiologists (ASA) physical status classification I-III;
4. Patients scheduled for elective laparoscopic gastrointestinal surgery;
5. Willingness to provide written informed consent and comply with the treatment regimen;
6. Absence of severe organic diseases, psychiatric disorders, or preoperative delirium.

Exclusion Criteria:

1. Preoperative Mini-Mental State Examination (MMSE) score <20;
2. Electrocardiographic evidence of severe bradycardia (heart rate <50 beats per minute);
3. Presence of skin lesions or infections at the electrical stimulation site;
4. History of preoperative chemotherapy or radiotherapy;
5. Concomitant severe organic diseases with compromised tolerance to interventions;
6. Prior exposure to Transcutaneous Electrical Acupoint Stimulation (TEAS) or transcutaneous auricular vagus nerve stimulation (taVNS) with documented insensitivity;
7. Inability to communicate normally, dementia, hearing impairment, or severe psychiatric disorders.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | The first to third days after surgery
  Whether delirium occurred after surgery（by 3D-CAM）

SECONDARY OUTCOMES:
IL-6 andTNF-α level | before operation（Before anesthesia），the end of the operation（Immediately after the sewing is finished）
  the level of IL-6 andTNF-α in the participant's serum（by ELISA）
VAS pain score | The first to third days after surgery
  Assessed with a VAS score scale, the highest is 10 and the lowest is 0, the higher the more severe the pain
Early activities | Post-operative period until discharge（in about a week）
  The first time to be able to get out of bed and move
Time to first postoperative anal defecation | Post-operative period until discharge（In about a week）
  Time to first postoperative anal defecation
Adverse events | The first to third days after surgery
  Nausea and vomiting, sore throat, itching

CONTACTS AND LOCATIONS:
Overall Officials: Lulu Ji, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The IPDs collected in the experiment were published only as the results of the paper